CLINICAL TRIAL: NCT04312048
Title: the Effect of Vaginal Isosorbide Mononitrate Administration in Reducing Pain During Cooper Intrauterine Device Insertion in Nulliparous Women : a Randomized Controlled Trial
Brief Title: the Effect of Isosorbide Mononitrate in Reducing Pain During Cooper Intrauterine Device Insertion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Samy aly ashour, assistant professor obstetrics and gynecology, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 00249
Record Dates: First submitted 2020-03-14; First posted 2020-03-18 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: IUD Insertion Pain
MeSH Terms: interventions — isosorbide-5-mononitrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isosorbide Mononitrate (Experimental): one tablet of Isosorbide Mononitrate (40 mg) vaginally 3 hours prior to copper IUD insertion
  Interventions: Drug: Isosorbide mononitrate
- placebo (Placebo Comparator): one tablet of placebo vaginally 3 hours prior to copper IUD insertion
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Isosorbide mononitrate — one tablet of Isosorbide Mononitrate (40 mg) vaginally 3 hours prior to copper IUD insertion
  Arms: Isosorbide Mononitrate
Drug: placebo — one tablet of placebo vaginally 3 hours prior to copper IUD insertion
  Arms: placebo

SUMMARY:
The aim of the study is to evaluate the efficacy of isosorbide mononitrate vaginal administration in reducing pain during copper IUD insertion in nulliparous women

ELIGIBILITY:
Inclusion Criteria:

* nulliparous women requesting copper IUD device insertion

Exclusion Criteria:

* parous women, contraindications to IUD insertion, allergy or contraindication to isosorbide mononitrate, uterine anomaly

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-10-25 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
pain during IUD insertion | 5 minutes
  intensity of patient-perceived pain at time of IUD insertion, using a visual analog scale. The VAS scale is graded from 0 to 100 on a 100 mm horizontal straight line, where 'zero' corresponds to no pain at all, and '100' to the worst possible pain imaginable.

SECONDARY OUTCOMES:
duration of IUD insertion | 5 minutes
  duration of IUD insertion from speculum in to speculum out

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud alalfy, MD, Principal Investigator — Cairo University
Locations (1):
- Ahmed Samy, Giza, Egypt